CLINICAL TRIAL: NCT01627197
Title: Adjuvant Intraarterial Chemotherapy Following Surgery in Treating Patients with Locally Advanced Bladder Cancer
Brief Title: Adjuvant Intraarterial Chemotherapy Following Surgery to Treat Locally Advanced Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Chair of Urology, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012009; 2012009 (Other: Sun Yat-sen University Clinical Research 5010 Program)
Record Dates: First submitted 2012-06-13; First posted 2012-06-25 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer
Keywords: Effects of Chemotherapy; intraarterial chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Intraaterial chemotherapy (Active Comparator): This is an open-label, prospective, multicenter, randomized, controlled phase 3 two-arm study.Patients with locally advanced TCC of the bladder are randomized to 1 of 2 treatment arms
  Arm 1 (treatment):'Surgery of percutaneous catheter system for arterial chemotherapy is done in the Department of Invasive Technology. All medications were administered using percutaneous catheter system via a modified Seldinger technique.Gemcitabine 800 mg/m2 intra-arterial,cisplatin 25 mg/m2 intra-arterial once a week for 3 weeks followed by 1-week rest period. Maximum of 3 cycles. Treatment begins between 1-5 weeks after radical operation (within 40 days is recommended).
  Interventions: Procedure: Surgery of percutaneous catheter system
- Watchful waiting (No Intervention): Arm 2 (control): No immediate post-surgery treatment. Patients undergo observation followed by cisplatin and gemcitabine as in arm I at local relapse, or receive intravenously chemotherapy with cisplatin and gemcitabine at multiple metastases

INTERVENTIONS:
Procedure: Surgery of percutaneous catheter system — Intraarterial (IA) catheterization was done in the Department of Invasive Technology. All medications were administered using percutaneous catheter system via a modified Seldinger technique. An angiographic catheter was inserted through the femoral artery into the internal iliac artery. The catheter tips were located superior to the origin of bilateral common artery.
  Arms: Intraaterial chemotherapy

SUMMARY:
Effect of adjuvant intra-arterial chemotherapy to control tumor progression in patients cystectomized for locally advanced bladder cancer.

DETAILED DESCRIPTION:
For locally advanced bladder cancer patients, tumor relapse rates after radial cystectomy were even as high as 50%-62%.Five-year disease-specific survival and OS rates in the organ-confined disease (defined as ≤pT3a) were 78.9% and 68%, respectively. For the non-organ-confined disease (defined as pT3b or higher), the rates were about 36.8% and 30.3%, respectively.Systemic chemotherapy can only prolong survival for up to 14.8 months, although with multiple severe adverse effects, such as neutrocytopenia, infection/sepsis, renal dysfunction, mucositis, or gastrointestinal toxicity. Additionally, the mortality rate associated with systemic chemotherapy was about 1%-4%.Therefore, the objective of our study was to determine if adjuvant intra-arterial chemotherapy with GC was able to reduce the systemic drug toxicities and yield a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed localized invasive bladder cancer following standardize radical cystectomy.
* Transitional cell carcinoma of bladder, stage pT3-4,N1-3,M0.Transitional cell carcinoma may be with or without squamous cell carcinoma and/or adenocarcinoma components.
* Male or female, 18 years of age or older, estimated life expectancy ≥ 6 months.
* ECOG performance status 0 or 1.
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase[SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normal (ULN).Total serum bilirubin≤ 1.5 x upper limit of normal (ULN).
* Absolute neutrophil count (ANC) ≥ 1500/μL
* Platelets ≥ 75,000/μL
* Hemoglobin ≥ 8.0 g/dL
* White blood cell count ≥ 3500/μL
* Creatinine clearance rate,Ccr ≥ 40ml/min
* Cardiac function level 0~2.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests,and other study procedures.

Exclusion Criteria:

* Bladder cancer without any transitional cell carcinoma component,such as adenocarcinoma,squamous cell carcinoma,small cell carcinoma
* Evidence of distant metastasis beyond the pelvis.
* No definitely pathological stage,such as no pathologic examination of perivesical fat,unable to differentiate pT2 and pT3,not performing lymph node dissection or regional lymph nodes cannot be assessed as the dissected lymph node number is less than ten.
* Prior neoadjuvant chemotherapy (systemic or intra-arterial) three months preoperatively, not including intra-vesical infusion chemotherapy.
* Prior pelvic radiation therapy dosage ≥ 30Gy six months preoperatively.
* Serious liver and kidney dysfunction.
* Accompanied with other serious diseases.
* Severe/unstable angina, arrhythmia,symptomatic heart failure, hypertension that cannot be controlled by medications and 6 months for myocardial infarction.
* Non-compliance of regular follow-up due to psychological, social, family and geographical and other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
recurrence free survival rate | 60 months

SECONDARY OUTCOMES:
overall survival | 60 months
Cancer specific survival | 60 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Jian Zhou, M.D Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes